CLINICAL TRIAL: NCT05582005
Title: An Observational Study of Emergence and Hypoactive Delirium After Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gianluca Bertolizio, MD, FRCPC, Associate Professor, Anesthesiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2023-9181
Record Dates: First submitted 2022-10-03; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Emergence Delirium; Hypoactive Delirium; Pain
MeSH Terms: conditions — Emergence Delirium; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: noninvasive blood pressure, 3 lead ECG, peripheral oxygen saturation — Children 3 year old and younger, scheduled for elective MRI, that are not intubated or require higher oxygen support and with no parents/guardians refusal will be placed on an electrocardiogram during post-anesthesia recovery. The NIPE monitor will be connected to the patients monitor in the PACU. Values will be recorded from the time of patient awaking until the patient meets the discharge criteria from PACU not before 1 hour.

SUMMARY:
Early postoperative negative behaviour (ePONB), such as pain, emergence delirium (ED) and hypoactive delirium, is a relevant clinical problem during recovery from anesthesia. Specifically, many children often present with different forms of negative behavior namely ED, hypoactive delirium or pain. Such negative behavior differs in terms of evolution, treatment, prognosis and clinical implications. Furthermore, there is overlap between tools used to measurement postoperative pain and ED. As a result, the assessment of the different forms of negative behavior are often compromised by the presence of postoperative pain. Therefore, the application of scales used to measure negative behaviour in postanesthetic, non-surgical patients aged 3 years and under scheduled for elective MRI may clarify the presence of ED, hypoactive delirium and pain. An improved understating of postanesthetic negative behavior is important in order to help implement appropriate measures so as to better treat these patients.

DETAILED DESCRIPTION:
The restless recovery from anesthesia is a relevant clinical problem that can be present in up to 80% of surgical cases. The incidence varies with age, anesthetic agents, type of surgery, and definition of the children behavior.

Unsettle behavior after anesthesia is associated with patient injury, damage to incision sites, exacerbated parental anxiety, increased nursing workload and cost of the healthcare system. Moreover, agitated children are seven times more likely to have new-onset separation anxiety, apathy, eating and sleeping problems.

The term early postoperative negative behavior (e-PONB) includes different unsettle behaviors after awakening and differentiates early phase from later postoperative behavioral changes. The more relevant components of e-PONB have been identified as pain and Emergence Delirium (ED).

ED a mental disturbance during the recovery from general anesthesia consisting in hallucinations, delusions and confusion manifested by moaning, restlessness, involuntary physical activity, and thrashing in bed. ED occurs within the first 20 min of recovery from anesthesia and often lasts 5-15 minutes and is self-limited.

The five-item Pediatric Anesthesia Emergence Delirium (PAED) scale is the gold standard to assess ED in the pediatric population. However, the diagnosis of ED may be affected by the concurrent presence postsurgical pain. A recent investigation found that only three of the five items of the PAED are delirium-specific ('Eye contact, 'Awareness of the surroundings', 'Purposeful actions'), whereas the other two ('Restlessness' and 'Inconsolability') are noted. As a consequence, if the child has 'no eye contact' and is 'no aware of surroundings,' emergence delirium should be suspected. On the contrary, a child showing 'Abnormal facial expression,' 'Crying' and being 'Inconsolable,' likely suffers of pain. The ED I and II score have been defined as the sum of the first 3-item (eye contact, purposeful movement, and awareness of surrounding) and the last 2-item scores (restlessness and inconsolability) of the PAED scale, respectively.

In up to 15% of children, however, the discrimination between ED and Pain remains impossible. In nonverbal children, in fact, pain is routinely assessed with the Face, Legs, Activity, Cry, Consolability (FLACC) scale. The PAED scale and the FLACC scale overlap on three items ('Inconsolability', 'Purposeful actions' and 'Restlessness'), which may lead to misdiagnose pain or ED.

Moreover, one in four children suffering from ED can present with a hypoactive delirium. Children are quiet, confused and disoriented: they do not make eye contact with the caregiver and may not be aware of their surroundings. Rather than being restless, agitated, and making non-purposeful movements, these children would only make minimal movements when awake, are non-communicative, and do not respond to social interactions. Primarily described in intensive care, hypoactive delirium is less recognized during the emergence from general anesthesia. In children, the Cornell Assessment of Pediatric Delirium (CAP-D) revise scale has been proposed to diagnose hypoactive delirium, but data are limited to one study on postsurgical patients.

In order to properly investigate ED and hypoactive delirium without the interference of concomitant pain, studies should be performed in a context of general anesthesia without any painful interventions. Children receiving general anesthesia for Magnetic Resonance Imaging (MRI) represent the ideal population free of "nociceptive stimulation" to investigate the incidence of ED and hypoactive delirium. However, up to one third of preschool children recovering from general anesthesia after MRI studies may show a FLACC score compatible with pain. Children experiencing ED were three times more likely to be also scored with pain.

In conclusion, children awaking from anesthesia might present different forms of negative behavior after anesthesia, namely ED, hypoactive delirium or pain. The evolution, treatment, prognosis and clinical implications of these conditions are different. There is a real practical need for a bedside tool to differentiate pain, ED and hypoactive delirium.

More recently, heart rate variability (HRV) has been proposed as a surrogate measure of pain and distress. In fact, HRV is affected by the balance between sympathetic and parasympathetic tone, and the high frequency changes of HRV is primarily mediated by and specific to the parasympathetic nervous system. The phenomena of pain, fear, anxiety and intraoperative nociception have proven to be accompanied by changes in HRV1.

The newborn infant parasympathetic evaluation (NIPE) is a non-invasive, standardized continuous measurement of HRV. The cardiac signal is extrapolated from the electrocardiogram and respiratory rate (RR) series are computed between two heart beats, resampled at 8 Hz, mean centered and normalized over a 64-second moving window. A wavelet based high pass filter over 0.15 Hz is applied in order to keep parasympathetic related variations only, which are mainly influenced by the respiratory cycle. The NIPE monitor displays two averaged measurements: the average NIPE (NIPEa) results from the average of NIPE measured over the previous 20 minutes, and current NIPE (NIPEc) results from the average of NIPE measured over the previous 64 seconds. A non-disclosed algorithm derived from the high frequency changes of the HRV calculates a score between 0 and 100, where a score of 0 indicates minimal parasympathetic tone and maximal nociception and a score of 100 indicates maximal parasympathetic tone and minimal nociception. To date, NIPE has shown promising results in the assessment of pain and neonatal comfort. In a recent study performed in postsurgical children at the Montreal Children's Hospital, the NIPE showed a significant correlation with pain but not with ED. Although the explanation remains speculative, it is possible that a some of the criteria of PAED are noyt associated with a variation of the parasympathetic tone (and therefore NIPE).

Should these results be confirmed, NIPE might be helpful to rule out the presence of pain and exclude ED.

ELIGIBILITY:
Inclusion Criteria:

* Children ≤ 3 years old, scheduled for elective MRI.
* Patients whose parents are fluent in French or English.

Exclusion Criteria:

* Intubated patients or have higher oxygen requirements
* Parent/guardian refusal

As this study will be conducted with only one NIPE monitor, and it will be devoted to the patient for about 1 hours, two consecutive patients cannot be enrolled in the study. In this case, the second patient will be considered eligible but excluded, and data will not be collected.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preschool Children
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Post-anesthesia negative behaviors (pain, emergence delirium and hypoactive delirium) | 1 hour
  Validation of NIPE as a tool to predict and assess post-anesthesia negative behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada